CLINICAL TRIAL: NCT01299194
Title: A Randomised Controlled Trial of Atorvastatin as an Anti-Inflammatory Agent in Non-Cystic Fibrosis Bronchiectasis in Patients With Pseudomonas Aeruginosa
Brief Title: Atorvastatin in Bronchiectasis in Patients With Pseudomonas Aeruginosa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-022042-24
Record Dates: First submitted 2010-10-21; First posted 2011-02-18 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: BRONCHIECTASIS
Keywords: BRONCHIECTASIS; PSEUDOMONAS AERUGINOSA; STATIN; OUTCOME
MeSH Terms: conditions — Bronchiectasis; Pseudomonas Infections | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATORVASTATIN (Active Comparator): Atorvastatin 80mg once daily for 3 months, 1.5 month wash out, then Placebo for 3 months
  Interventions: Drug: ATORVASTATIN
- PLACEBO (Placebo Comparator): Placebo 3 months, then washout for 1.5 months, then Atorvastatin 80mg once daily
  Interventions: Drug: ATORVASTATIN

INTERVENTIONS:
Drug: ATORVASTATIN — 80mg once daily for 3 months

SUMMARY:
Statins are a class of drug used to prevent heart attacks and strokes by lowering blood cholesterol levels. They have also been found to have a beneficial "side effect" of lowering the level of inflammation in the body. This is thought to be one of the reasons they are effective in treating heart attacks and strokes. Laboratory experiments have shown that statins reduce lung inflammation in response to bacteria and this is a promising development for the treatment of chest infections.

Bronchiectasis is a chronic disabling lung disease characterised by chronic sputum production and recurrent chest infections. 2/3 of patients are chronically colonised with bacteria (normally the lungs are sterile) and this leads inflammation in the lung and in the rest of the body.

There are no effective treatments for bronchiectasis other than antibiotics for chest infections. With increasing antibiotic use, there is increasing antibiotic resistance and new treatments for this disease are needed.

The investigators intend to study Atorvastatin in patients with bronchiectasis with colonization with pseudomonas aeruginosa. The investigators will give Atorvastatin to 16 patients with this disease while 16 patients will receive placebo. This will be a crossover study where patients will receive atorvastatin or placebo for 3 months, followed by a statin wash out period of 6 weeks. Thereafter the groups will cross over and the group receiving atorvastatin will now receive placebo and those receiving placebo will receive atorvastatin for 3 months. The investigators will measure inflammation in their lungs and in the rest of their body before and after treatment with atorvastatin. The investigators will also assess their quality of life and number of chest infections over a 7.5 month period.

This pilot study will determine if there is any role for statins are an anti-inflammatory agent in patients with bronchiectasis.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONAL FOR STUDY Bronchiectasis is a chronic debilitating respiratory condition. Patients suffer daily cough, excess sputum production and recurrent chest infections because of inflamed and permanently damaged airways. It is a common with a Scottish incidence of 1 in 1,000 to 1 in 10,000. Over 600 patients in Edinburgh are monitored in secondary care. They frequently utilise primary and secondary care resources through consultations, A&E attendances and inpatient admissions. The economic burden is huge- hospital admissions alone for bronchiectasis cost NHS Lothian just over 1 million pounds alone last year.

LIMITATIONS OF TREATMENT There are few evidence based long term treatments currently available. Long term antibiotics are a feasible option, but with the increasing problems of antimicrobial resistance and side effects, in particular Clostridium difficile and methicillin resistant Staphylococcus aureus (MRSA), there is an international drive to reduce antibiotic usage. There is an urgent need for novel non antibiotic treatments.

Statins as a potential new non antibiotic treatment in bronchiectasis Excessive neutrophilic airways inflammation is the central feature of bronchiectasis. This paradoxically both promotes bacterial colonisation and perpetuates damage to the airways creating a vicious cycle of bacterial colonisation and inflammation.1-3

Statins have been shown to have powerful anti-inflammatory effects.4-6 In animal models, statins can reduce neutrophil recruitment to the inflamed lung and reduce protease activity.7 Statin treatment has been shown to reduce epithelial cell adherence and invasion by Streptococcus pneumoniae in-vitro suggesting a role for statins in preventing bacterial colonisation.8 In healthy controls exposed to lipopolysaccharide to induce acute lung inflammation, pre-treatment with simvastatin reduced neutrophil accumulation in the lung and inhibited production of myeloperoxidase, tumour necrosis factor-alpha, matrix metalloproteinases and C-reactive protein.9 There was also an increase in neutrophil apoptosis, suggesting that statins may aid the resolution of inflammation in the airway.10

STUDY HYPOTHESIS We hypothesise that long term statin treatment will improve patients' symptoms through its anti-inflammatory effect. The beneficial effects on patient symptoms (cough, sputum volume, bacterial load, airway function, exercise tolerance, exacerbation frequency and health related quality of life) will be consequent on reduced neutrophilic airways inflammation.

Planned study

* This is a randomised double blind placebo controlled cross over trial to assess the efficacy of atorvastatin therapy in patients with clinically significant bronchiectasis.
* No such study has previously been undertaken (PUBMED Search "statins" and "bronchiectasis" 18 March 2010- no relevant articles).
* This is a unique proof of principle study assessing a new non antibiotic treatment that could benefit all patients with clinically significant bronchiectasis, without the side effect profile of long term antibiotics.
* Following this proof of principle study, we aim to design a large multi-centred study assessing long term statins as a new treatment.

  1. Stockley RA et al. Elastolytic activity of sputum and its relation to purulence and to lung function in patients with bronchiectasis. Thorax 1984;39(6):408-413.
  2. Hill AT et al. Association between airway bacterial load and markers of airway inflammation in patients with stable chronic bronchitis. Am J Med 2000;109(4):288-95.
  3. Inflammation: a two-edged sword-the model of bronchiectasis. Cole PJ. Eur J Respir Dis Suppl. 1986;147:6-15.
  4. Ridker PM et al. C-reactive protein levels and outcomes after statin therapy. N Engl J Med 2005;352:20-8.
  5. Terblanche M et al. Statins and Sepsis: multiple modifications at multiple levels. Lancet Infect Dis. 2007; 7(5):358-368.
  6. Vaughan CJ, Murphy MB, Buckley BM. Statins do more than just lower cholesterol. Lancet 1996;348:1079-82.
  7. Fessler MB et al. A role for HMG coenzyme A reductase in pulmonary inflammation and host defense. Am J Respir Crit Care Med 2005;171:606-15.
  8. Rosch JW et al. Statins protect against fulminant pneumococcal infection and cytolysin toxicity in a mouse model of sickle cell disease. J Clin Invest 2010; 120(2);627-35.
  9. Shyamsundar M et al. Simvastatin decreases lipopolysacchraide-induced pulmonary inflammation in healthy volunteers. Am J Respir Crit Care Med. 2009 179:1107-1114.
  10. Watt AP et al. Neutrophil apoptosis, proinflammatory mediators and cell counts in bronchiectasis. Thorax 2004;59(3):231-6.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 will be recruited.
* All will have an established radiological diagnosis of bronchiectasis (CT of the chest).
* Patients colonised with Pseudomonas Aeruginosa.
* Able to give informed consent.

Exclusion Criteria:

* Current smokers or ex-smokers of less than 1 year; >15 pack year history
* Cystic fibrosis
* Active allergic bronchopulmonary aspergillosis
* Active tuberculosis
* Poorly controlled asthma
* Pregnancy or breast feeding
* Known allergy to statins
* Active malignancy
* Chronic liver disease
* Established cardiovascular or cerebrovascular disease
* Statin use in the last year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-11; Primary Completion 2015-06 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is a reduction in cough at 3 months compared to baseline as measured by the Leicester Cough Questionnaire score. | 7.5 months

SECONDARY OUTCOMES:
pulmonary physiology and assessment of exercise capacity | 7.5 months
24 hour sputum volume | 7.5 months
qualitative and quantitative bacteriology | 7.5 months
health related quality of life and health care utilisation | 7.5 months
exacerbation frequency | 7.5 months
safety of statin therapy | 7.5 months
Airways and systemic inflammation | 7.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam T Hill, MBChB MD, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Bedi P, Chalmers JD, Graham C, Clarke A, Donaldson S, Doherty C, Govan JRW, Davidson DJ, Rossi AG, Hill AT. A Randomized Controlled Trial of Atorvastatin in Patients With Bronchiectasis Infected With Pseudomonas Aeruginosa: A Proof of Concept Study. Chest. 2017 Aug;152(2):368-378. doi: 10.1016/j.chest.2017.05.017. Epub 2017 May 26. PMID 28554732